CLINICAL TRIAL: NCT01636440
Title: Reliability of Measuring Conditioned Pain Modulation With the Nociceptive Withdrawal Reflex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Aalborg University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 070/12; SNF: SPUM 33CM30_124117
Record Dates: First submitted 2012-07-05; First posted 2012-07-10 (Estimated); Last update posted 2013-01-21 (Estimated); Status verified 2013-01

CONDITIONS: Healthy Volunteers
Keywords: Conditioned Pain Modulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Reliability (Other): The same testing procedure is repeated after a delay of 7 days to test the reliability of the measure
  Interventions: Device: Conditioned Pain Modulation

INTERVENTIONS:
Device: Conditioned Pain Modulation — Measure of the conditioned pain modulation with the nociceptive withdrawal reflex and ice water stimulation
Device: Conditioned Pain Modulation — Suprathreshold electrical stimulation with 1.5 times the mean electrical pain detection threshold

SUMMARY:
Conditioned pain modulation is the ability of the spine to describe changes in pain perception, if two different painful stimulations take place. The reliability of the conditioned pain modulation has not been studied, the instruments used to measure the conditioned pain modulation are sparse and have proven difficult to use in a well reproductible way. This study is using an existing pain test, relying on the reflex in a muscle after a painful electrical stimulation. We will test 34 healthy volunteers in order to test the reliability of the conditioned pain modulation with the nociceptive withdrawal reflex combined to a ice water test.

DETAILED DESCRIPTION:
Background

Chronic pain is characterized by changes in the central processing of sensory inputs. Quantitative sensory tests (QST) explore central excitability in humans and have the potential to detect altered central pain processing in individual patients.

QST were developed to assess the responses to sensory stimuli for research purposes, providing psychophysical and electrophysiological methods for the assessment of the nociceptive system. Reliability is an essential condition for using QST in research and clinical practice. It can be defined as the consistency of measurements across time, patients or observers, and the extent to which it is error-free. Three categories have been assessed for reliability in QST measures: intra-rater, inter-rater and test-retest reliability. Reliability of QST measures in healthy volunteers are encouraging in regard to good repeatability of QST measures over the time in the same subjects. Inter-rater reliability, a prerequisite to compare different measures in between different studies, are also highly encouraging.

Under normal conditions, pain after application of a test nociceptive stimulus is attenuated by the application of an additional "conditioning" noxious stimulus to a remote body region, reflecting diffuse endogenous inhibition. This is defined as conditioned pain modulation (CPM), also known as the "pain inhibits pain" paradigm. CPM has been object of much work in the last years. It goes back to the exploration of endogenous analgesia via descending pain-modulatory systems, which started about three decades ago in animal models. Descending inhibitory pathways are under cerebral control, mediating modulation of pain perception by emotional, motivational and cognitive factors. Alterations of CPM are a known risk factor concerning acute and chronic pain syndromes.

Very few reliability studies on CPM have been conducted to date. To our knowledge, only S. Cathcart et al used occlusion cuff algometry and pressure pain detection to assess the test-retest reliability in healthy volunteers. A study in chronic pain patients from our group has shown great variability in CPM. It is unclear whether this phenomenon is related to high interindividual variability of the CPM measure itself, or to poor reliability. In an analysis of own data extracted from a pharmacological study, CPM measured at three different sessions in patients with low back pain displayed very poor reliability.

The nociceptive withdrawal reflex is an electrophysiological measure. Compared to psychophysical measures which rely on the subject's pain perception, the reflex could be a more reproducible and stable measure over time.

Objective

The primary aim of the present study is to assess the reliability of CPM using the nociceptive withdrawal reflex as test stimulus and the ice water test as conditioning stimulus in 34 consecutive patients, with a 7 days interval between two sessions.

Secondary aim is to compare the reliability of CPM with the nociceptive withdrawal reflex to the reliability of CPM assessed with subjective pain assessments, i.e. pain threshold and pain intensity after electrical stimulation.

Methods

Repeated assessments of CPM using the nociceptive withdrawal reflex threshold, electrical pain detection threshold and suprathreshold electrical stimulation of the skin, with ice-water as conditioning stimuli in all three models. There will be a 7 days interval between two measurements.

ELIGIBILITY:
Inclusion Criteria:

* Male Gender
* Age 18-65
* Signed Informed Consent

Exclusion Criteria

* Signs or suspicion of neurologic dysfunction or disease
* Ongoing treatment with any drug known to influence pain modulation: any analgesic, antidepressant, anticonvulsant or benzodiazepine
* Intake of any analgesic drug during the 48h preceding the experiment.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2012-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Reliability of CPM with the nociceptive withdrawal reflex | two minutes after the cold pressor test

SECONDARY OUTCOMES:
Reliability of CPM with electric pain detection threshold | two minutes after the cold pressor test
Reliability of CPM with suprathreshold electrical pain detection threshold stimulation | two minutes after the cold pressor test

CONTACTS AND LOCATIONS:
Overall Officials: Michele Curatolo, MD, Study Director — University Hosptial Bern
Locations (1):
- Dep. of Anesthesiology and Pain Medicine, Bern University Hospital, Bern, Switzerland

REFERENCES:
- [Derived] Biurrun Manresa JA, Fritsche R, Vuilleumier PH, Oehler C, Morch CD, Arendt-Nielsen L, Andersen OK, Curatolo M. Is the conditioned pain modulation paradigm reliable? A test-retest assessment using the nociceptive withdrawal reflex. PLoS One. 2014 Jun 20;9(6):e100241. doi: 10.1371/journal.pone.0100241. eCollection 2014. PMID 24950186